CLINICAL TRIAL: NCT03441906
Title: QUEST: QUality of Life and Experiences of Sarcoma Trajectories
Acronym: QUEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-3881
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2019-03

CONDITIONS: Quality of Life; Sarcoma; Diagnostic Interval; Diagnostic Pathway; Care Needs
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

The prognosis of patients with rare cancers in general and sarcomas in particular suffers from delay in diagnosis. Routes to diagnosis for sarcoma need to be quicker and more streamlined, but have neither been studied in detail in larger numbers before, nor in a direct comparison between two countries with different health systems. Comprehensive assessment of diagnostic delays and its determinants, including demographic, clinical, psychosocial and health care system factors, is necessary to improve referral pathways and come to best practice and patient reported outcomes for sarcoma patients.

Research questions to be answered:

This study aims to quantify diagnostic delay (including patient, general practitioner and system delay) and evaluates routes to diagnosis and referral to sarcoma expert centres in the Netherlands and England; to comprehensively evaluate risk factors of diagnostic delay; determine the association between diagnostic delay and outcomes (health-related quality of life, quality-adjusted life years, patient satisfaction, TNM classification, time to local/distant relapse and overall survival); and to assess differences between both countries. This should lead to advices about faster referral where possible.

DETAILED DESCRIPTION:
The researchers will conduct a longitudinal cohort study among all sarcoma patients (≥18 years of age) that will be newly diagnosed in 1.5 years period from October 1st 2017 to March 30st 2019 in one of the participating study centers (5 centers in The Netherlands, 3 centers in England).

Patients will be invited before the start of treatment (with a two months eligibility window) and receive a questionnaire on diagnostic delay, risk factors and patient-reported outcomes. The questionnaire on patient-reported outcomes will be completed again 3 months, 6 months, 1-year and 2 years later.

Data collection will be done within PROFILES, an international registry for cancer patient reported outcomes (www.profilesregistry.nl). Clinical data will be collected through cancer registries and the junior investigator will collect extra data from patients' records.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis ≥ 18 years
* Diagnosis of sarcoma (histology confirmed by sarcoma histopathologist; according to ICD-10-GM codes C40 and C41 for bone sarcoma and C49 for soft-tissue sarcoma)
* Able to communicate in English (or Dutch)
* Mental capacity to provide informed consent and to participate in the study (as determined by the referring health care professional)
* Patients must be able to complete questionnaires themselves
* Patients must be under treatment or follow-up at one of the participating hospitals.

Exclusion Criteria:

* Too ill to complete questionnaires (according to advice from (former) treating specialist)
* Patients with desmoids fibromatosis will be excluded because of the non-malignancy of the disease; and patients with gastrointestinal stromal tumours (GIST; ICD-10-GM codes C15-20, C26, C48 and C80) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with sarcoma, see inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Baseline
  Health-related quality of life

SECONDARY OUTCOMES:
Diagnostic interval | Relationship between diagnostic interval and quality of life at baseline
  Time to diagnosis
Factors influencing diagnostic interval | At baseline
  Risk factors to experience a long diagnostic interval
QALY | Baseline
  Quality adjusted life years
Psychologic impact | 2 years
  several measures will be taken into account, such as HADS etc
Change in quality of life | 2 years
  Change in QoL throughout follow up
PFS | through study completion, an average of 2 years
  progression free survival
OS | Through study completion, an average of 2 years
  Overall survival
Change in QALY | Change from baseline throughout follow-up of 2 years
  Quality adjusted life years

CONTACTS AND LOCATIONS:
Overall Officials: Winette van der Graaf, Prof, MD, Principal Investigator — Radboud University Medical Center
Locations (8):
- Netherlands (5):
  - NKI-AVL, Amsterdam
  - UMCG, Groningen
  - LUMC, Leiden
  - Radboudumc, Nijmegen
  - Erasmus medical centre, Rotterdam
- United Kingdom (3):
  - Royal Orthopaedic Hospital, Birmingham
  - Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soomers V, Desar IM, van de Poll-Franse LV, Husson O, van der Graaf WT. Quality of life and experiences of sarcoma trajectories (the QUEST study): protocol for an international observational cohort study on diagnostic pathways of sarcoma patients. BMJ Open. 2020 Oct 26;10(10):e039309. doi: 10.1136/bmjopen-2020-039309. PMID 33109665